CLINICAL TRIAL: NCT05477108
Title: A Phase I, Randomized, Double-blind, Single-dose, Partial Replicate, 3-way Cross-over Study to Assess the Lung Exposure Bioequivalence of Budesonide, Glycopyrronium, and Formoterol Delivered by BGF MDI HFO Compared With BGF MDI HFA
Brief Title: Study to Assess the Lung Exposure Bioequivalence of Budesonide, Glycopyrronium, and Formoterol Delivered by BGF MDI With Next-Generation Propellant Compared With BGF MDI With HFA Propellant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5985C00005; 118313 (Other: IND No)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Corticosteroid; Long acting muscarine agonist (LAMA); Long acting beta agonist; Propellant; Bioequivalence; Lung exposure; Healthy subjects; Inhaled corticosteroid (ICS); Long-acting β2 agonist (LABA); Next generation propellant (NGP)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Charcoal; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: BGF MDI HFO 160/7.2/4.8 μg ex-actuator with oral activated charcoal (Experimental): Subjects will receive Test formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA. The reference formulation will be administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
  Interventions: Drug: Treatment A (BGF MDI HFO with oral activated charcoal); Drug: Treatment B (BGF MDI HFA with oral activated charcoal)
- Treatment B: BGF MDI HFA 160/7.2/4.8 μg ex-actuator with oral activated charcoal (Experimental): Subjects will receive Reference formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA. The reference formulation will be administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
  Interventions: Drug: Treatment A (BGF MDI HFO with oral activated charcoal); Drug: Treatment B (BGF MDI HFA with oral activated charcoal)

INTERVENTIONS:
Drug: Treatment A (BGF MDI HFO with oral activated charcoal) — Subject will receive 4 inhalations as a single dose with oral activated charcoal - test formulation; administered during 1 Treatment Period.
  Other Names: Budesonide / Glycopyronium / Formoterol fumarate pressurized inhalation suspension, HFO
Drug: Treatment B (BGF MDI HFA with oral activated charcoal) — Subject will received 4 inhalations as a single dose with oral activated charcoal - reference formulation; administered during 2 Treatment Periods.
  Other Names: Budesonide / Glycopyronium / Formoterol fumarate pressurized inhalation suspension, HFA

SUMMARY:
The study will assess the Pharmacokinetic (PK) and safety of BGF MDI [Budesonide/glycopyrronium/formoterol (BGF) metered dose inhaler (MDI)] formulated with 2 different propellants :Hydrofluoroolefin (HFO) and Hydrofluoroalkane (HFA) with oral activated charcoal in healthy subjects (male or female).

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, single-dose, single-center, partial-replicate, 3 way cross-over study.

The study will comprise:

* Screening period: up to 28 days prior to first dosing;
* Three treatment periods : Subject will be resident in the Clinical Unit from the morning on the day before dosing with BGF MDI (Day 1 of Treatment Period 1), until 24 hours following the final dose (Day 2 of Treatment Period 3 a washout period of 3 to 7 days between each dose;
* Follow-up: Within 3 to 7 days after the last administration of BGF MDI.

Subjects will receive 3 single-dose treatments of BGF MDI [Test formulation Treatment A (BGF MDI HFO); Reference formulation Treatment B (BGF MDI HFA)] on Day 1 of each Treatment Period (1, 2, and 3) following an overnight fast of at least 8 hours. There will be a washout period of 3 to 7 days between each dose.

Each subjects will be involved in the study for up to 55 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male and/or female subjects aged 18 - 60 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating, confirmed at screening.
* Have a Body Mass Index (BMI) between 18 and 35 kg/m2 inclusive and weigh at least 50 kg and no more than 120 kg inclusive.
* Subjects must have a Forced expiratory volume in the first second (FEV1) ≥ 80% of the predicted normal value and an FEV1/FVC (Forced vital capacity) > 70% regarding age, height, and ethnicity at the screening visit.
* Subjects must demonstrate proper inhalation technique and have the ability to properly use an MDI device after training.
* Provision of signed and dated, written informed consent prior to any study specific procedures.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational Medicinal Product (IMP).
* History of narrow angle glaucoma not adequately treated and/or change in vision that may be relevant.
* History of symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention.
* Unresectable cancer that has not been in complete remission for at least 5 years.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.
* Any clinically significant abnormal findings in physical examination, or vital signs at screening.
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and HIV antibody.
* Subject has a positive RT-PCR test for SARS-CoV-2 prior to randomization.
* Subject has clinical signs and symptoms consistent with SARS-CoV-2 infection, eg, fever, dry cough, dyspnea, sore throat, fatigue, or laboratory confirmed acute infection with SARS-CoV-2.
* Subject who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated, Intensive Care Unit stay).
* Recent (within 14 days prior to admission to the Clinical Unit) exposure to someone who has COVID-19 symptoms or tested positive for SARS-CoV-2.
* Has a current occupation that involves routine exposure to potential COVID-19 patients or sources of SARS-CoV-2 infection (eg, healthcare worker).
* History of any respiratory disorders such as asthma, COPD, or idiopathic pulmonary fibrosis.
* Known or suspected history of drug abuse.
* Receipt of any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to randomization
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to BGF.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within 3 months prior to screening.
* Positive screen for drugs of abuse or cotinine at screening or on admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day or would likely be unable to refrain from the use of caffeine-containing beverages during confinement.
* Subjects who have previously received BGF MDI HFO.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00005&attachmentIdentifier=e5c8ceb9-9dfe-4567-b720-c71a64fac7e1&fileName=d5985c00005-study-synopsis_final_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 29 July 2022 to 11 April 2023 at a single study center - Parexel Early Phase Clinical Unit (Baltimore).
Pre-assignment Details: The Screening period was up to 28 days. Informed Consent Form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment.
Groups:
- Treatment Sequence ABB: Participant received 3 single dose treatment of Budesonide, Glycopyrronium, Formoterol (BGF) Metered Dose Inhaler (MDI) in 3 occasions.
  Participant received BGF MDI Hydrofluoroolefin (HFO) (Treatment A); then BGF MDI Hydrofluoroalkane (HFA)(Treatment B); and then BGF MDI HFA (Treatment B) with oral activated charcoal prior and post dosing (A or B) on Day 1 with a washout period of 3 to 7 days between each dose.
- Treatment Sequence BAB: Participant received 3 single dose treatment of BGF MDI in 3 occasions. Participant received BGF MDI HFA (Treatment B); then BGF MDI HFO (Treatment A); and then BGF MDI HFA (Treatment B) with oral activated charcoal prior and post dosing (A or B) on Day 1 with a washout period of 3 to 7 days between each dose.
- Treatment Sequence BBA: Participant received 3 single dose treatment of BGF MDI in 3 occasions. Participant received BGF MDI HFA (Treatment B); then BGF MDI HFA (Treatment B); and then BGF MDI HFO (Treatment A) with oral activated charcoal prior and post dosing (A or B) on Day 1 with a washout period of 3 to 7 days between each dose.
Period: Overall Study
Arm/Group | Treatment Sequence ABB | Treatment Sequence BAB | Treatment Sequence BBA
Started | 36 | 36 | 36
Completed | 35 | 35 | 33
Not Completed | 1 | 1 | 3
Not completed — Participants randomized, not treated | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — withdrawn from study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Set consisted of all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABB | Treatment Sequence BAB | Treatment Sequence BBA | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (10.5) | 37.8 (11.7) | 38.6 (11.1) | 38.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 17 | 46
  Male | 22 | 21 | 19 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 24 | 19 | 64
  White | 12 | 10 | 13 | 35
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma (Peak) Drug Concentration (Cmax )
Description: Bioequivalence (Cmax) of the lung exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO compared with BGF MDI HFA was assessed.
Time Frame: Pre-dose, 2 minutes, 5 minutes,10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hours (h), 2 h, 4 h, 8 h, 12h and 24 hours post-dose on Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: The PK analysis set consisted of all randomized participants who had at least 1 primary PK parameter that could be calculated, and who had no important protocol deviations thought to impact on the analysis of the PK data. Here, number of participants analyzed refers to number analyzed for each specific outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Groups:
- Treatment A: Subjects received BGF MDI HFO; 4 inhalations as a single dose with oral activated charcoal, test formulation.
- Treatment B (Replicate 1); Treatment B (Replicate 2): Subjects received BGF MDI HFA; 4 inhalations as a single dose with oral activated.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 97 | 99
picograms per milliliter (pg/mL)
  Budesonide | 1078 (61.09) | 1111 (63.42) | 1045 (73.36)
  Glycopyrronium: number analyzed (Participants) | 97 | 95 | 90
  Glycopyrronium | 14.31 (98.78) | 15.22 (96.13) | 15.17 (92.85)
  Formoterol: number analyzed (Participants) | 100 | 97 | 99
  Formoterol | 18.82 (75.45) | 19.31 (74.53) | 19.35 (80.39)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Budesonide Pharmacokinetic Parameters (US approach); Test type: Equivalence — For Cmax, the intra-participant CV% in Treatment B (reference arm) was 42.91. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.1028 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 104.24, 90% CI 2-sided [95.78 to 113.44] — Geometric mean ratio is calculated as A/B
Statistical Analysis 2: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Glycopyrronium Pharmacokinetic Parameters (US approach); Test type: Equivalence — For Cmax, the intra-participant CV% in Treatment B (reference arm) was 40.85. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.0831 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 93.45, 90% CI 2-sided [84.31 to 103.58] — Geometric mean ratio is calculated as A/B
Statistical Analysis 3: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Formoterol Pharmacokinetic Parameters (US approach); Test type: Equivalence — For Cmax, the intra-participant CV% in Treatment B (reference arm) was 40.66. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.0971 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 100.14, 90% CI 2-sided [91.90 to 109.11] — Geometric mean ratio is calculated as A/B
Statistical Analysis 4: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Budesonide Pharmacokinetic Parameters (EU approach); Test type: Equivalence — For Cmax, the analysis was conducted using an analysis of variance including fixed effects for treatment, sequence, period and subject within sequence. The PK parameter was log-transformed prior to analysis. The intra-participant CV% in Treatment B (reference arm) was 42.66. Bioequivalence was concluded since the 90% CI for the geometric mean ratio were within the expanded equivalence limits of 73.29% to 136.44% and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 103.12, 90% CI 2-sided [94.44 to 112.60] — Geometric mean ratio is calculated as A/B
Statistical Analysis 5: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Glycopyrronium Pharmacokinetic Parameters (EU approach); Test type: Equivalence — For Cmax, the analysis was conducted using an analysis of variance including fixed effects for treatment, sequence, period and subject within sequence. The PK parameter was log-transformed prior to analysis. The intra-participant CV% in Treatment B (reference arm) was 40.75. Bioequivalence was concluded since the 90% CI for the geometric mean ratio were within the expanded equivalence limits of 74.24% to 134.70% and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 93.39, 90% CI 2-sided [85.29 to 102.26] — Geometric mean ratio is calculated as A/B
Statistical Analysis 6: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Formoterol Pharmacokinetic Parameters (EU approach); Test type: Equivalence — For Cmax, the analysis was conducted using an analysis of variance including fixed effects for treatment, sequence, period and subject within sequence. The PK parameter was log-transformed prior to analysis. The intra-participant CV% in Treatment B (reference arm) was 40.81. Bioequivalence was concluded since the 90% CI for the geometric mean ratio were within the expanded equivalence limits of 74.21% to 134.75% and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 99.70, 90% CI 2-sided [91.44 to 108.71] — Geometric mean ratio is calculated as A/B

2. Primary Outcome: Area Under Plasma Concentration Time Curve From Zero to Infinity (AUCinf)
Description: Bioequivalence (AUCinf) of the lung exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO compared with BGF MDI HFA was assessed.
Time Frame: Pre-dose, 2 minutes, 5 minutes,10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h, 12 h and 24 hours post-dose on Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)*pg/mL
Groups:
- Treatment A: Subjects received BGF MDI HFO 160/7.2/4.8 μg per actuation; 4 inhalations as a single dose with oral activated charcoal, test formulation.
- Treatment B (Replicate 1): Subjects received BGF MDI HFA 160/7.2/4.8 μg per actuation; 4 inhalations as a single dose with oral activated.
- Treatment B (Replicate 2): Subjects received BGF MDI HFA per actuation; 4 inhalations as a single dose with oral activated.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
hour (h)*pg/mL
  Budesonide | 2533 (61.57) | 2479 (61.34) | 2507 (76.08)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 45.66 (245.3) | 33.60 (223.9) | 64.50 (271.8)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 54.12 (85.90) | 53.36 (85.09) | 53.70 (111.9)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Budesonide Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUCinf, the intra-participant CV% in Treatment B (reference arm) was 34.29. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.0593 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 107.76, 90% CI 2-sided [100.35 to 115.72] — Geometric mean ratio is calculated as A/B
Statistical Analysis 2: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Glycopyrronium Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUCinf, the intra-participant CV% in Treatment B (reference arm) was 86.08. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.2925 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Ratio Mean (%) = 112.22, 90% CI 2-sided [92.27 to 136.49] — Geometric mean ratio is calculated as A/B
Statistical Analysis 3: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Formoterol Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUCinf, the intra-participant CV% in Treatment B (reference arm) was 47.07. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.1250 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 101.45, 90% CI 2-sided [91.76 to 112.15] — Geometric mean ratio is calculated as A/B

3. Primary Outcome: Area Under the Plasma Concentration Curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: Bioequivalence (AUClast) of the lung exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO compared with BGF MDI HFA was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)*pg/mL
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 97 | 99
hours (h)*pg/mL
  Budesonide | 2460 (63.25) | 2398 (62.89) | 2421 (78.43)
  Glycopyrronium: number analyzed (Participants) | 97 | 95 | 90
  Glycopyrronium | 25.11 (182.1) | 20.34 (190.9) | 34.58 (180.3)
  Formoterol: number analyzed (Participants) | 100 | 97 | 99
  Formoterol | 36.47 (112.8) | 35.68 (117.6) | 35.83 (160.9)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Budesonide Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUClast, the intra-participant CV% in Treatment B (reference arm) was 35.68. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.0668 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 106.87, 90% CI 2-sided [99.30 to 115.01] — Geometric mean ratio is calculated as A/B
Statistical Analysis 2: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Glycopyrronium Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUClast, the intra-participant CV% in Treatment B (reference arm) was 74.17. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.2735 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 102.02, 90% CI 2-sided [89.12 to 116.79] — Geometric mean ratio is calculated as A/B
Statistical Analysis 3: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Formoterol Pharmacokinetic Parameters (US approach); Test type: Equivalence — For AUClast, the intra-participant CV% in Treatment B (reference arm) was 66.88. An analysis was conducted based on the RSABE method for a partial-replicate 3-way cross-over design. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since criteria bound was -0.2210 (<0) and point estimate for geometric mean ratio was within 80% and 125%; Geometric Mean Ratio (%) = 107.76, 90% CI 2-sided [94.91 to 122.36] — Geometric mean ratio is calculated as A/B
Statistical Analysis 4: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Budesonide Pharmacokinetic Parameters (EU approach); Test type: Equivalence — For AUClast, the analysis was conducted using an analysis of variance including fixed effects for treatment, sequence, period and subject within sequence. The PK parameter was log-transformed prior to analysis. Bioequivalence was concluded since the 90% CI for the geometric mean ratio were fully contained within the predefined equivalence limits of 80% to 125%; Geometric Mean ratio (%) = 106.10, 90% CI 2-sided [98.39 to 114.41] — Geometric mean ratio is calculated as A/B
Statistical Analysis 5: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Glycopyrronium Pharmacokinetic Parameters (EU approach); Test type: Equivalence — [test comment as in outcome 3, analysis 4]; Geometric Mean Ratio (%) = 97.02, 90% CI 2-sided [84.18 to 111.82] — Geometric mean ratio is calculated as A/B
Statistical Analysis 6: Comparison: Treatment A vs Treatment B (Replicate 1) vs Treatment B (Replicate 2); Statistical Comparison of Key Formoterol Pharmacokinetic Parameters (EU approach); Test type: Equivalence — [test comment as in outcome 3, analysis 4]; Geometric Mean Ratio (%) = 105.74, 90% CI 2-sided [92.59 to 120.75] — Geometric mean ratio is calculated as A/B

4. Secondary Outcome: Time to Reach Peak or Maximum Observed Concentration or Response Following Drug Administration (Tmax)
Description: The tmax as PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Treatment B (Replicate 1): Subjects received BGF MDI HFA 160/7.2/4.8 μg per actuation; 4 inhalations as a single dose with oral activated. A partial-replicate design was used in which the reference treatment was administered on 2 occasions to assess within-participant variability and widen the 90% CI limits charcoal, reference formulation.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 97 | 99
hours
  Budesonide | 0.33 [0.07 to 1.13] | 0.32 [0.07 to 4.00] | 0.33 [0.05 to 1.02]
  Glycopyrronium: number analyzed (Participants) | 97 | 95 | 90
  Glycopyrronium | 0.05 [0.03 to 0.33] | 0.07 [0.03 to 0.22] | 0.05 [0.03 to 0.20]
  Formoterol: number analyzed (Participants) | 100 | 97 | 99
  Formoterol | 0.08 [0.03 to 0.22] | 0.08 [0.03 to 0.22] | 0.08 [0.03 to 0.20]

5. Secondary Outcome: Half Life Associated With Terminal Slope (λz) of a Semi Logarithmic Concentration Time Curve (t½λz)
Description: The t½λz as PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
hours
  Budesonide | 3.661 (32.13) | 3.304 (30.86) | 3.656 (33.60)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 9.063 (300.9) | 6.025 (308.2) | 13.30 (302.7)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 6.997 (53.32) | 6.444 (64.95) | 7.082 (77.98)

6. Secondary Outcome: Terminal Rate Constant (λz)
Description: The λz PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
1/hour
  Budesonide | 0.1893 (32.13) | 0.2098 (30.86) | 0.1896 (33.60)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 0.07648 (300.9) | 0.1151 (308.2) | 0.05213 (302.7)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 0.09907 (53.32) | 0.1076 (64.95) | 0.09787 (77.98)

7. Secondary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation From Zero to Infinity (MRTinf)
Description: The MRTinf PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
hours
  Budesonide | 3.893 (21.04) | 3.771 (23.43) | 3.978 (22.85)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 12.04 (294.9) | 7.991 (295.0) | 18.30 (293.0)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 9.139 (51.58) | 8.497 (62.87) | 9.254 (75.92)

8. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F)
Description: The CL/F PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/hour (L/h)
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
Litre/hour (L/h)
  Budesonide | 250.7 (61.57) | 258.2 (61.34) | 255.2 (76.08)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 630.7 (245.3) | 857.2 (223.9) | 446.5 (271.8)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 354.8 (85.90) | 359.8 (85.09) | 357.5 (111.9)

9. Secondary Outcome: Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Based on Terminal Phase) (Vz/F)
Description: The Vz/F PK profiles of BGF administered as BGF MDI HFO and BGF MDI HFA with oral activated charcoal was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 101 | 96 | 99
Litre (L)
  Budesonide | 1324 (57.12) | 1231 (59.34) | 1346 (69.25)
  Glycopyrronium: number analyzed (Participants) | 89 | 90 | 73
  Glycopyrronium | 8247 (41.09) | 7451 (53.30) | 8566 (44.65)
  Formoterol: number analyzed (Participants) | 99 | 94 | 98
  Formoterol | 3581 (49.08) | 3345 (49.90) | 3653 (46.55)

10. Secondary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of single doses of BGF MDI HFO and BGF MDI HFA with oral activated charcoal in healthy subjects was assessed.
Time Frame: From screening (Day -28 to Day -1) up to 55 days
Population: The safety analysis set included all participants who received at least 1 inhalation of any BGF MDI.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 103 | 105 | 104
Participants
  Any AE | 12 | 19 | 4
  Any SAE | 0 | 0 | 0
  Any SAE with outcome of death | 0 | 0 | 0
  Any AE leading to discontinuation of study intervention | 0 | 0 | 0
  Any possibly related AE | 4 | 6 | 2
  Any possibly related SAE | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to Day -1) up to 55 days
Description: The safety analysis set included all participants who received at least 1 inhalation of any BGF MDI.
  Adverse events that were collected from the start of screening throughout the Treatment period up to and including the final follow-up Phone call was presented.
Groups:
- Treatment B (Replicate 1): Subjects received BGF MDI HFA per actuation; 4 inhalations as a single dose with oral activated.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/105 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/105 | 0/104
Other Adverse Events (participants affected / at risk) | 12/103 | 19/105 | 4/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=103) | Treatment B (Replicate 1) (N=105) | Treatment B (Replicate 2) (N=104)
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 2 | 2 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 1 | 1 | 0
Vessel puncture site swelling (General disorders) | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT05477108/Prot_SAP_000.pdf